CLINICAL TRIAL: NCT03365037
Title: Study of Therapeutic Effect of Electret Static Physiotherapy Film on Acute Soft Tissue Closed Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Yichong, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH20121030A
Record Dates: First submitted 2017-11-25; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Soft Tissue Injuries
MeSH Terms: conditions — Soft Tissue Injuries | interventions — Polypropylenes

STUDY DESIGN:
Intervention Model Description: A randomized, open, parallel controlled, non inferiority clinical trial design was used in this trial.Objective to evaluate the safety and effectiveness of electret static physiotherapy film in Beijing Youshilin science and Technology Development Co., Ltd.The patients were followed up after receiving the electret static physiotherapy film, and the treatment and complication rate of the patients were observed after the electret static physiotherapy film was attached to the patient.The data were compared between the experimental group and the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electret electrostatic physiotherapyFilm (Experimental): Patients with acute soft tissue injury treated with electret electrostatic physiotherapyFilm
  Interventions: Drug: Electret electrostatic physiotherapyFilm
- Fracture healing film (Active Comparator): Patients with acute soft tissue injury treated with fracture healing film
  Interventions: Drug: Fracture healing film

INTERVENTIONS:
Drug: Electret electrostatic physiotherapyFilm — Patients with acute soft tissue injury treated with electret electrostatic physiotherapyFilm
  Other Names: polypropylene
  Arms: Electret electrostatic physiotherapyFilm
Drug: Fracture healing film — Patients with acute soft tissue injury treated with Fracture healing film
  Other Names: Teflon,2011-2640661
  Arms: Fracture healing film

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of electret static physiotherapy film developed by Beijing Youshilin science and Technology Development Co., Ltd., to treat acute soft tissue injury by sticking to the affected area

DETAILED DESCRIPTION:
Design of randomized, open, parallel controlled non inferiority clinical trial.A total of 60 patients were included in the trial, including 30 subjects in the experimental group and 30 subjects in the control group. The experimental disease was acute soft tissue closed injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute soft tissue injury diagnosed by Western Medicine
* Ability to communicate well with the researcher and comply with the requirements of the validation
* Participants agreed to participate in the clinical validation and follow the validation program requirements, and signed the informed consent form

Exclusion Criteria:

* There are important organs (heart and lung) serious disease history, or have autoimmune disease history, such as rheumatism, SLE, or have a history of immune dysfunction, such as suffering from aids
* Patients with cardiac pacemaker
* Patients with open wounds
* Pregnant and lactating women
* Patients with history of mental illness
* Participants participated in other medical device trials or drug clinical trials within three months
* The researchers believe that the participants who are not eligible for clinical validation should be considered
* Patients who need to be treated with drugs
* Patients requiring physical therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

PRIMARY OUTCOMES:
Number of cured persons | 7 days after treatment (±2 days)
  Pain, swelling, bruising and other symptoms and signs of integration to reduce more than 95%, the normal joint movement

SECONDARY OUTCOMES:
Number of adverse events | 7 days after treatment (±2 days)
  allergic skin rash

CONTACTS AND LOCATIONS:
Overall Officials: Peixun Zhang, Doctor, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided